CLINICAL TRIAL: NCT05657080
Title: An Investigation on Cytosponge and Molecular Biomarkers to Identify Patients With Gastric Intestinal Metaplasia (GIM)
Brief Title: Cytosponge for Gastric Intestinal Metaplasia
Acronym: CyGIM
Status: Recruiting | Type: Observational
Sponsor: University of Cambridge (Other)
Collaborators: University College London Hospitals (Other); Nottingham University Hospitals NHS Trust (Other)
Responsible Party: Principal Investigator, Massimiliano di Pietro, MD, Senior Clinical Investigator Scientist, University of Cambridge
Other Study IDs: CyGIM_v1
Record Dates: First submitted 2022-11-30; First posted 2022-12-20 (Actual); Last update posted 2024-05-08 (Actual); Status verified 2024-05

CONDITIONS: Gastric Cancer; Gastric Intestinal Metaplasia; Gastric Atrophy
Keywords: early cancer detection; gastric premalignant lesions; non-invasive cancer screening
MeSH Terms: conditions — Stomach Neoplasms; Gastritis, Atrophic | interventions — Endoscopy, Digestive System; Blood Specimen Collection

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Human tissue obtained in this study will include:
  1. Upper gastrointestinal tract tissue from endoscopic biopsy samples for the purpose of tissue diagnosis and for discovery validation of molecular biomarkers
  2. Blood
  3. Gastric juice (via Cytosponge [as supernatant] or via endoscopic aspiration)
  4. Gastric cytology (via Cytosponge)
  Nucleic acids (DNA/RNA) will be extracted from tissue biopsies, gastric juice vesicles and blood.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (2):
- Cases: This will include patients with:
  * existing diagnosis of proximal GIM undergoing endoscopic surveillance
  * a new diagnosis of proximal GIM requiring repeat endoscopy
  * a historical diagnosis of GIM retrieved from the pathology records through retrospective analysis and lost in follow up
  * gastric adenocarcinoma from upper GI multidisciplinary meeting.
  Interventions: Device: Cytosponge-TFF3
- Controls: Controls will be patients with no known premalignant conditions of the upper GI tract and fit to undergo an upper endoscopy. They will be recruited via standard referral routes for upper GI endoscopy due to upper GI symptoms via standard referral routes. Individuals must be able to provide informed consent.
  Interventions: Device: Cytosponge-TFF3

INTERVENTIONS:
Device: Cytosponge-TFF3 — Cytosponge is a less invasive procedure than endoscopy and consists of an expandable, spherical mesh, which is attached to a string and contained within a soluble capsule. Five minutes after swallowing (once the capsule has dissolved), the spherical mesh, which measures around 3cm in diameter can be retrieved by pulling on the string. Upon retrieval the Cytosponge scrapes against the surface of the top of the stomach and oesophagus and collect epithelial cells. The Cytosponge sample is then placed into a preservative fluid and the specimen is processed for molecular tests. Trefoil Factor 3 (TFF3) is a protein that is expressed in intestinal type epithelia of the gastrointestinal tract. TFF3 is the best biomarker, which can be coupled to the Cytosponge to diagnose intestinal metaplasia.
  Other Names: Upper GI endoscopy; Blood sampling

SUMMARY:
Gastric cancer has a very poor prognosis. The disease is often diagnosed at a late stage, when curative treatment options are limited or ineffective. There is a condition that predisposes to gastric cancer, known in medical terms as Gastric intestinal metaplasia (GIM). This pre-cancerous condition can be diagnosed with an endoscopic camera test, but it often very subtle and can be missed at routine endoscopy. There is evidence that about 7% of gastric cancers are missed at previous endoscopy.

The Cytosponge-trefoil factor 3 (TFF-3) is a pill on a string combined to a molecular biomarker which could help early diagnosis of gastric cancer and GIM. Cytosponge-TFF3 has been showed in previous research to be useful to diagnose Barrett's oesophagus, a condition of the food pipe similar to GIM.

The aim of this study is to investigate the utility of the Cytosponge in combination with molecular biomakers to diagnose GIM

DETAILED DESCRIPTION:
This is a case-control study whose goal is to compare the non-endoscopic test (Cytosponge-TFF3) to standard endoscopy to diagnose gastric intestinal metaplasia (GIM), a precursor lesion for gastric cancer. The main objective of the study is to determine the sensitivity and specificity of the Cytosponge-TFF3 to detect gastric intestinal metaplasia (GIM) affecting the proximal stomach.

In parallel to this clinical study, a experimental study will be carried out aimed at evaluating the utility of molecular biomarkers to refine/improve the diagnostic accuracy of the Cytosponge test. The hypothesis is that the non-invasive Cytosponge, in combination with molecular biomarkers, can accurately detect GIM to the same extent as conventional, but more invasive, endoscopic procedures.

Patients will be invited to participate in the study if they are due their surveillance endoscopy, because they have the disease of interest (GIM or GC; cases) or have been referred for an upper endoscopy for abdominal complaint (controls). On the day of the endoscopy the patient will swallow the Cytosponge under supervision of a trained research nurse prior to the endoscopic procedure. The participant will also provide information on demographics, clinical exposures (alcohol, tobacco, drugs), have measurements of weight and height taken and they will also complete a validated gastrointestinal symptoms questionnaire. A blood sample will be taken from the cannula used for the sedatives or through venepuncture. The patients will then undergo their planned endoscopy with additional sampling of gastric juice (suctioned through the endoscope) and some additional research biopsies in addition to a standardized clinical protocol to diagnose GIM. The above research procedures will be performed prior and during the endoscopy. No further research procedures will follow afterwards beyond the day of the endoscopy.

The aim is to develop a non-invasive test which can be used to screen patients at risk for GIM to allow early detection and treatment of pre-cancerous gastric lesions and ultimately reduce the number of patients dying of gastric cancer.

ELIGIBILITY:
Inclusion Criteria:

* Any participant 18 years and above clinically fit for an endoscopy with GIM of the proximal stomach confirmed on previous biopsies or gastric adenocarcinoma of intestinal type (cases)
* Any participant 18 years and above clinically fit for an endoscopy with upper GI symptoms leading to referral for endoscopy (controls)
* Ability to provide informed consent

Exclusion Criteria:

* Individuals with a diagnosis of an oro-pharynx, oesophageal or gastro-oesophageal tumour (T2 staging and above), or symptoms of dysphagia.
* Patients with previous diagnosis of Barrett's oesophagus oesophageal varices, stricture or requiring dilatation of the oesophagus.
* Patients unable to stop anticoagulation therapy/medication timely before the procedure (heparin or tinzaparin, apixaban, rivaroxaban, dabigatran, edoxaban; 48 hours, warfarin; 5 days, clopidogrel; 7 days)
* Individuals who have had a myocardial infarction or any cardiac event less than six months ago.
* Individuals who have had a cerebrovascular event < 6 months ago where their swallowing has been affected
* Patients who have had previous treatments such as Photodynamic therapy (PDT), Radiofrequency ablation or Argon Plasma Coagulation for dysplastic Barrett's oesophagus
* Participants who are unable to provide informed consent.
* Participants under age 18.

NB - Endoscopy is generally avoided in pregnant women and therefore it is unlikely that any pregnant women will be included although pregnancy would not be an absolute contraindication. Pregnancy/ pregnancy test will not be recorded as part of the trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Cases and controls will be treated in the UK.
  Cases:
  * Patients with an existing diagnosis of proximal GIM referred for endoscopic surveillance will
  * Patients with newly diagnosed GIM who require a repeat endoscopy for complete endoscopy biopsy mapping.
  * Patients with a historical diagnosis of GIM retrieved from the pathology records and in need of endoscopic surveillance based on clinical guidelines.
  * Patients with gastric cancer (intestinal type) recruited from the multidisciplinary team meeting and undergoing endoscopy and laparoscopy as part of their regular cancer staging or surveillance.
  Controls will be referred from primary or secondary care with upper GI symptoms and no known premalignant conditions of the upper GI tract.
Sampling Method: Non-Probability Sample
Enrollment: 226 (Estimated)
Dates: Start 2023-10-16 (Actual); Primary Completion 2024-09-30 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Sensitivity of Cytosponge for GIM | 2 months
  Proportion of GIM cases extending to the proximal stomach diagnosed based on gold standard endoscopy with biopsies correclty classified by Cytosponge-TFF3 testing

SECONDARY OUTCOMES:
Histopathological disease stage | through study completion, an average of 1 year
  A panel of clinical and molecular biomakers on biopsies, Cytosponge and blood, will be used to construct a model to predict the histopathological stage of disease (OLGA/OLGIM + grade of neoplasia)
Number of participants with device-related adverse events as assessed by CTCAE v4.0 | 2 weeks from recruitment
  Adverse events realted to Cytosponge will be recorded immediate after administration and at 2 weeks after study visit

CONTACTS AND LOCATIONS:
Overall Officials: Massimiliano di Pietro, MD, Principal Investigator — University of Cambridge; Andreas Hadjicinolaou, MD PhD, Study Director — University of Cambridge
Locations (1):
- Cambridge Clinical Research Centre, Cambridge, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided
Patient details will be pseudo-anonymised, with no identifiable information to be shared outside the clinical research team. Electronic transfers of pseudo-anonymised data will meet industry and NHS-mandated standards including encryption to at least Advanced Encryption Standard (AES) 256. Data will be stored on study database for 10 yrs after study completion, in a linked anonymised manner. Participants will be aware that their PID might be accessed by external regulatory bodies for the purposes of assessing legal compliance and meeting relevant regulatory obligations. Anonymised clinical and lifestyle information may be transferred and stored in international repositories for access by international researchers in line with patient consent.
  Temporary access to PID might occur in the event of pathology review by central pathology panel, but PID will not be stored outside local research institution.

REFERENCES:
- [Background] Banks M, Graham D, Jansen M, Gotoda T, Coda S, di Pietro M, Uedo N, Bhandari P, Pritchard DM, Kuipers EJ, Rodriguez-Justo M, Novelli MR, Ragunath K, Shepherd N, Dinis-Ribeiro M. British Society of Gastroenterology guidelines on the diagnosis and management of patients at risk of gastric adenocarcinoma. Gut. 2019 Sep;68(9):1545-1575. doi: 10.1136/gutjnl-2018-318126. Epub 2019 Jul 5. PMID 31278206
- [Background] Pimentel-Nunes P, Libanio D, Marcos-Pinto R, Areia M, Leja M, Esposito G, Garrido M, Kikuste I, Megraud F, Matysiak-Budnik T, Annibale B, Dumonceau JM, Barros R, Flejou JF, Carneiro F, van Hooft JE, Kuipers EJ, Dinis-Ribeiro M. Management of epithelial precancerous conditions and lesions in the stomach (MAPS II): European Society of Gastrointestinal Endoscopy (ESGE), European Helicobacter and Microbiota Study Group (EHMSG), European Society of Pathology (ESP), and Sociedade Portuguesa de Endoscopia Digestiva (SPED) guideline update 2019. Endoscopy. 2019 Apr;51(4):365-388. doi: 10.1055/a-0859-1883. Epub 2019 Mar 6. PMID 30841008
- [Background] Fitzgerald RC, di Pietro M, O'Donovan M, Maroni R, Muldrew B, Debiram-Beecham I, Gehrung M, Offman J, Tripathi M, Smith SG, Aigret B, Walter FM, Rubin G; BEST3 Trial team; Sasieni P. Cytosponge-trefoil factor 3 versus usual care to identify Barrett's oesophagus in a primary care setting: a multicentre, pragmatic, randomised controlled trial. Lancet. 2020 Aug 1;396(10247):333-344. doi: 10.1016/S0140-6736(20)31099-0. PMID 32738955
- [Background] Ross-Innes CS, Debiram-Beecham I, O'Donovan M, Walker E, Varghese S, Lao-Sirieix P, Lovat L, Griffin M, Ragunath K, Haidry R, Sami SS, Kaye P, Novelli M, Disep B, Ostler R, Aigret B, North BV, Bhandari P, Haycock A, Morris D, Attwood S, Dhar A, Rees C, Rutter MD, Sasieni PD, Fitzgerald RC; BEST2 Study Group. Evaluation of a minimally invasive cell sampling device coupled with assessment of trefoil factor 3 expression for diagnosing Barrett's esophagus: a multi-center case-control study. PLoS Med. 2015 Jan 29;12(1):e1001780. doi: 10.1371/journal.pmed.1001780. eCollection 2015 Jan. PMID 25634542
- [Background] Hadjinicolaou AV, Azizi AA, O'Donovan M, Debiram I, Fitzgerald RC, Di Pietro M. Cytosponge-TFF3 Testing can Detect Precancerous Mucosal Changes of the Stomach. Clin Gastroenterol Hepatol. 2022 Jun;20(6):1411-1412. doi: 10.1016/j.cgh.2021.07.047. Epub 2021 Aug 3. PMID 34358719
- [Background] Cui L, Zhang X, Ye G, Zheng T, Song H, Deng H, Xiao B, Xia T, Yu X, Le Y, Guo J. Gastric juice MicroRNAs as potential biomarkers for the screening of gastric cancer. Cancer. 2013 May 1;119(9):1618-26. doi: 10.1002/cncr.27903. Epub 2013 Jan 18. PMID 23335180
- [Background] Ikeda F, Shikata K, Hata J, Fukuhara M, Hirakawa Y, Ohara T, Mukai N, Nagata M, Yoshida D, Yonemoto K, Esaki M, Kitazono T, Kiyohara Y, Ninomiya T. Combination of Helicobacter pylori Antibody and Serum Pepsinogen as a Good Predictive Tool of Gastric Cancer Incidence: 20-Year Prospective Data From the Hisayama Study. J Epidemiol. 2016 Dec 5;26(12):629-636. doi: 10.2188/jea.JE20150258. Epub 2016 Jun 4. PMID 27265836
- [Background] Gawron AJ, Shah SC, Altayar O, Davitkov P, Morgan D, Turner K, Mustafa RA. AGA Technical Review on Gastric Intestinal Metaplasia-Natural History and Clinical Outcomes. Gastroenterology. 2020 Feb;158(3):705-731.e5. doi: 10.1053/j.gastro.2019.12.001. Epub 2019 Dec 6. No abstract available. PMID 31816300